CLINICAL TRIAL: NCT07074119
Title: Sensor-Based Optimization of Therapy for Parkinson's Disease Patients With Motor Fluctuations
Acronym: SO-TOP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: NS-PARK Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: APHP180609; 2019-A00322-55 (Other: ANSM)
Record Dates: First submitted 2025-06-26; First posted 2025-07-20 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease (PD)
Keywords: Adjusment Therapy; Dyskinesis; Time ON; Time OFF; Bradykinesia; Parkinson Kinetic Graff; Body-worn Sensors; Parkinson Watch; self-reported diary
MeSH Terms: conditions — Parkinson Disease; Dyskinesias; Hypokinesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients of the control group will undergo the same protocol as patients in the experimental arm. However, data extracted from the BWS will be made available to the neurologist.
  Interventions: Device: wearable-based adjustment therapy
- Control group (Active Comparator): Patients of the control group will undergo the same protocol as patients in the experimental arm. However, data extracted from the BWS will be blinded and NOT be made available to the neurologist.
  Interventions: Device: wearable-based adjustment therapy

INTERVENTIONS:
Device: wearable-based adjustment therapy — * Patients will wear the BWS for 7 days prior to each of the visit : baseline (V1) at week 0, V2 at week 4 (phone call at 1 month), V3 at week 12 (3 months visit) and V4 at week 24 (6 months).
  * Data extracted from each session of monitoring with the BWS will be made available to the neurologist (only in the experimental group) prior to V1 (W0), V2 (W4), V3 (W12) and V4 (W24) respectively
  * Treatment adjustment will be guided by the current consensus guidelines for treatment adjustment for motor fluctuations in PD using reports from BWS data. Reports will be screened by neurologists before the patient's visit so the groups blinding is correctly observed

SUMMARY:
Although numerous tools have been developed in recent years with the enhancement of new technologies precision and the reduction of their size, still few medical devices are used in clinical routine in Parkinson's Disease. Knowledge about Parkinson's Disease motor symptoms has been widely improved especially thanks to objective monitoring of movements. However, patients are mostly observed in defined environment during scripted activities, which is per se distinct from the real life conditions. Besides, experts may agree on the limitations of the diary that is supposed to reflect the patient's status at home, while outpatients' visits may also not correctly enable the neurologist to catch up the everyday life condition of the patient. In order to overcome some of these issues, we hypothesize that the implementation of body-worn sensors at home monitoring could provide promising solutions. Yet, important information is missing: there is no previous randomized trial studying the additional value of body-worn sensors to improve motor symptoms, quality of life and ability to perform everyday life activities for example. To our knowledge, our study proposal is the first one to adjust therapy of patients with Parkinson's Disease based on the reports of body-worn sensors monitoring. If the efficacy and reliability of at home monitoring with sensors is proven, new healthcare guidelines could arise with the objective of a better and continuous patient's follow-up, remotely from the outpatient's visit.

DETAILED DESCRIPTION:
The study is Single Blind Randomized clinical trial. The participants are patients with Parkinson's Disease at the stage of motor fluctuations without dementia or levodopa-resistant axial symptoms who need therapeutic adjustments according to the neurologist opinion. The primary objectif is to assess the efficacy of the Body Worn Sensors (BWS)-based adjustment therapy, on add-on to usual care, on change in time spent in OFF state in PD patients with motor fluctuation requiring treatment adaptation. The primary endpoint is the change in daily time spent in OFF state between baseline and 6 months visit, measured as the mean daily time in OFF state upon 3 days on self-reported diary. Medical device under investigation, CE-marked (class IIA) under regulation UE 2017/745, is a body-worn sensor (BWS) that measures movements and analyses accelerometry data to report motor symptoms of Parkinson's Disease. The product is the PKG system (Global Kinetics Corporation, Melbourne Australia). This BWS embarks a dedicated algorithm that continuously reports severity scores of bradykinesia, dyskinesia and tremor over a week of monitoring. All the patients will wear the PKG Watch but results from BWS recording will be available for the neurologist to adapt the treatment, according to randomization allocation (Available in the experimental group only). In both groups (experimental and control group), the treatment will be adapted according to current guidelines. Four follow-up visits will be performed at M0 (W0), M1 (W4 +/- 7 days), M3 (W12 +/- 7 days) and M6 (W24 +/- 7 days) during outpatients clinics (except for M1 = phone call) where participants are usually followed. 13 centers in France participating to the NS-PARK network (French research Network for PD). The duration of recruitment will be 24 months. The duration of participation for each participant will be 6 months, the total duration of the study will be 31 months. For this study, 218 patients will be recruited.

ELIGIBILITY:
Inclusion criteria :

* Parkinson's since > 4 years
* Patient between years 46-83 (according to the BWS range of validity)
* Presence of motor fluctuations as defined by a score ≥ 2 (item 4.3) and a score ≥ 1 (item 4.4) of the MDS-UPDRS part IV
* At least 3 doses per day of L-Dopa
* Need of therapeutic adjustment because of motor fluctuations according to the neurologist opinion
* Hoehn and Yahr stage ≤ 3 in OFF state

Exclusion criteria :

* No signature of informed consent
* Anticipated uncompliance or inability to use the self-reported diary or to wear the devices
* Cognitive impairment (MMSE < 24)
* Patient treated with second line therapies ((Subcutaneous or digestive pump therapies or deep brain stimulation) or planed for the 6 next months.
* Pregnant or breastfeeding women
* Patients living in nursing home
* Patient already participating in another clinical investigation or interventional study.

Ages: 46 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Change in daily time spent in OFF state between baseline and 6 months visit, measured as the mean daily time in OFF state upon 3 days on self-reported diary. | Baseline (W0) and 6 months visit (W24)
  The daily time spent in OFF states will be reported by the patient on his/her diary per periods of thirty minutes each day for a duration of 3 days before baseline visit and before 6 months visit. For each day, the total daily time spent OFF will be calculated as the sum of every 30 minutes' periods stated as OFF time. This duration will be averaged over the 3 days period at baseline (W0 +/-7 days) and 6 months (W24 +/- 7 days) visits and the difference between the two visits will be calculated.

SECONDARY OUTCOMES:
Change in time spent in good ON state without troublesome dyskinesia (i.e. good time ON) between baseline and 6 months on self-reported diary (mean of previous 3 days) | Baseline (W0) and 6 months visits (W24)
  For each day, the total time spent in ON state without troublesome dyskinesia will be calculated as the sum of every 30 minutes periods stated as time spent in ON state without troublesome dyskinesia.
Change in time spent in ON state with troublesome dyskinesia between baseline and 6 months on self-reported diary (mean of previous 3 days) | baseline (W0) and 6 months visits (W24)
  For each day, the total time spent in ON state with troublesome dyskinesia will be calculated as the sum of every 30 minutes periods stated as time spent in ON state with troublesome dyskinesia in the diary. These durations will be averaged over the 3 days period at baseline (W0 +/- 7 days) and 6 months visits (W24 +/- 7 days) and the difference between the two visits will be calculated.
Change of Movement Disorder Society-Unified Parkinson's Disease Rating Scale part II (MDS-UPDRS part II-motor aspects of experiences of daily living) between baseline and 6 months | baseline (W0) and 6 months visits (W24)
  The Movement Disorder Society-Unified Parkinson's Disease Rating Scale part II (MDS-UPDRS part II ) score will be assessed at baseline and 6 months visits. The change will be calculated as the difference between the scores obtained at 6 months visit (W24 +/- 7 days) and baseline visit (W0 +/- 7 days).
  The minimum score of the MDS-UPDRS part II is 0 and the maximum score is 52, the higher score means a worse outcome.
Change of the score of Parkinson Disease Quality of life questionnaire (PDQ-39) related between baseline and 6 months | baseline (W0) and 6 months visits (W24)
  The Parkinson Disease Quality of life questionnaire (PDQ-39) is a self-questionnaire assessing disease related quality of life in PD. The patient will fill it in at baseline and 6 months visits. The change will be calculated as the difference between the scores obtained at 6 months visit (W24 +/- 7 days) and baseline visit (W0 +/- 7 days).
  The minimum score of the Parkinson Disease Quality of 0 and the maximum score is 156, the higher score means a worse outcome.
Number of patients with at least one dopaminergic drug-related side effects between groups during the study period. | baseline (W0), 1 month visit (W4), 3 months visit (W12) and 6 months (W24)
  Dopaminergic drug-related side effects will be collected at each visit: baseline (W0 +/- 7 days), phone call at 1 months (W4 +/- 7 days), 3 months visit (W12 +-/ 7 days), 6 months visit (W24 +/- 7 days). AE will be classified as related or not with anti-parkinsonian drug and rated according to their severity. The number and severity of anti-parkinsonian drug side effects will be compared across groups.
Number of patients with each type of Dopaminergic drug-related | baseline (W0), phone call at 2 months (W4 ), 3 months visit (W12 ), 6 months visit (W24)
  The side effects will be described in each group
Change of Movement Disorder Society-Unified Parkinson's Disease Rating Scale part I (MDS-UPDRS part I-non-motor aspects of experiences of daily living) between baseline and 6 months | baseline (W0) and 6 months visits (W24)
  Movement Disorder Society-Unified Parkinson's Disease Rating Scale part I (MDS-UPDRS part I) score will be assessed at baseline and 6 months visits. The change will be calculated as the difference between the scores obtained at 6 months visit (W24 +/- 7 days) and baseline visit (W0 +/- 7 days).
  The minimum score of the MDS-UPDRS part I is 0 and the maximum score is 52, the higher score means a worse outcome.
Changes in drug regimen during the study of Levodopa equivalent daily doses (LEDD) between baseline and 6 months | baseline (W0) and 6 months visit (W24)
  The change in LEDD between 6 months visit (V4) and baseline visit (V1) will be calculated as the difference.
Changes in drug regimens between baseline and 6 months | baseline (W0) and 6 months visits (W24)
  Antiparkinsonian and associated treatments will be systematically collected at baseline (W0 +/- 7 days) and 6 months (W24 +/- 7 days) visits. The number and type of changes (i.e. addition of drugs, discontinuation of drugs, increase / decrease of dosing) between baseline visit (W0) and 6 months visit (W24 +/- 7 days) will be described.
Number of consultations between baseline visit (W0) and 6 months visit | baseline (W0) and 6 months visits (W24)
  Number of consultations (general practitioner, neurologist, other specialist, advanced practice nurse) between baseline visit (W0) and 6 months visit (W24 +/- 7 days)
Number of hospitalization days between baseline visit (W0) and 6 months visit | baseline (W0) and 6 months visits (W24)

OTHER OUTCOMES:
Change in time spent in OFF state between baseline and 6 months based on the BWS assessment | baseline (W0) and 6 months visits (W24)
  It will be calculated on the basis of the BWS report according to the continuous monitoring of the patient during 7 days. OFF state periods are defined as time with BKS mild (25<BKS≤39.3 corresponding to BKS above the target range and below the 90th percentile of healthy controls) or BKS severe (39.3<BKS≤80, corresponding to BKS above the 90th percentile of healthy controls). Change will be calculated as the difference between values obtained at 6 months visit (W24 +/- 7 days) and baseline visit (W0 +/- 7 days).
Change in time spent in good ON state (i.e. time ON without troublesome dyskinesia) between baseline and 6 months based on the BWS assessment. | baseline (W0) and 6 months visits (W24)
  It will be calculated on the basis of the BWS report according to the continuous monitoring of the patient during 7 days. Time spent in ON state without troublesome dyskinesia will be defined as the sum of all 2' periods within the target range for BKS (BKS≤25) and below the 90th percentile for DKS (DKS≤47.2). Change will be calculated as the difference between values obtained at 6 months visit (W24 +/- 7 days) and baseline visit (W0 +/-7 days).
Change in time spent in ON state with troublesome dyskinesia between baseline and 6 months based on the BWS assessment | baseline (W0) and 6 months visits (W24)
  It will be calculated on the basis of the BWS report according to the continuous monitoring of the patient during 7 days. Time spent in ON state with troublesome dyskinesia will be defined as the sum of all 2 miutes periods BKS< 25 (normal range) and DKS>47.2 (above the 90th percentile). . Change will be calculated as the difference between values obtained at 6 months visit (W24 +/- 7 days) and baseline visit (W0 +/- 7 days).
Concordance of OFF state measure between the diary and the BWS reports | baseline (W0) and 6 months visits (W28)
  For each patient a concordance rate will be calculated as the number of 30 minutes' period (for all the visits with both diary and BWS assessments) rated as OFF in the diary and measures as OFF in the BWS report , divided by the number of 30 minutes' period rated as OFF in the diary. A period will be considered as OFF with the BWS report if the patient has BKS>25 during more than 50% of the non-immobile period (BKS≤80).
Concordance of the good time ON state (i.e. time ON without troublesome dyskinesia) between the diary and the BWS reports | baseline (W0) and 6 months visits (W24)
  For each patient a concordance rate will be calculated as the number of 30 minutes' period (for all the visits with both diary and BWS assessments) rated as good time ON in the diary and measures as good ON state in the BWS report, divided by the number of 30 minutes' period rated as good time ON in the diary. A period will be considered as good ON state with the BWS report if the patient has BKS≤25 and DKS≤47.2 during more than 50% of the non-immobile period (BKS≤80).
Concordance of the time ON state with troublesome dyskinesia in the diary and the time with dyskinesia given by the BWS report | baseline (W0) and 6 months visits (W24)
  For each patient a concordance rate will be calculated as the number of 30 minutes' period (for all the visits with both diary and BWS assessments) rated as time ON with troublesome dyskinesia in the diary and measures as time with dyskinesia in the BWS report, divided by the number of 30 minutes' period rated as time ON with troublesome dyskinesia in the diary.A period will be considered as ON state with troublesome dyskinesia with the BWS report if the patient has BKS ≤25 and DKS > 47.2 during more than 50% of the non-immobile period (BKS≤80).
The attractiveness of the Body Worn Sensor (BWS) from patients | 6 months visit (W24)
  The attractiveness will be assessed by scores of a user experience questionnaire System Usability Scale (SUS) at 6 months. The SUS will be filled-in separately by patients (in the 2 groups) at 6 months (W24+/- 7 days) visit.
The attractiveness of the Body Worn Sensor (BWS) from neurologists | 6 months visit (W24)
  The attractiveness will be assessed by scores of a user experience questionnaire System Usability Scale (SUS ) at 6 months. The SUS will be filled-in neurologists only in the BWS-based adjustment group.

CONTACTS AND LOCATIONS:
Overall Officials: David Grabli, Professor, Principal Investigator — Assistance Publique Hopitaux de Paris; Jean Chritophe Corvol, Professor, Study Director — Assistance Publique Hopitaux de Paris
Locations (1):
- Centre d'investigations cliniques Pitié-Salpêtrière University Hospital, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided